CLINICAL TRIAL: NCT01980498
Title: Multicenter Randomized Open Trial to Evaluate Efficacy of Fentanyl Pectin Nasal Spray vs Physician Choice-Usual Care in Reducing Predictable Breakthrough Pain at Swallowing in Head/Neck Cancer Patients Undergoing Radiotherapy
Brief Title: PEctin Rapid Fentanyl Efficacy Clinical Trial For pAin at Swallowing Undergoing radioTherapy
Acronym: PERFECT FAST
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: L.Molteni & C. dei F.lli Alitti-Soc. di Esercizio S.p.A. (Industry)
Collaborators: Consorzio Mario Negri Sud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOLT-2013-02; 2013-001271-20 (EudraCT Number)
Record Dates: First submitted 2013-10-21; First posted 2013-11-11 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2014-06

CONDITIONS: Predictable BTP at Swallowing in in Head/Neck Cancer Patients Undergoing Radiotherapy Already Receiving Opioid Therapy for Background Pain

ARMS (2):
- PecFent nasal spray (Experimental): Patients that have signed the ICF and met inclusion and exclusion criteria are randomly assigned 1:1 to receive one of the following IP-BTP treatments:
  1. Fentanyl pectin nasal spray (FPNS)
  2. Physician choice-Usual Care (PC-UC)
  Interventions: Drug: Fentanyl pectin nasal spray (FPNS)
- Physician choice-Usual Care (PC-UC) (Active Comparator): Patients that have signed the ICF and met inclusion and exclusion criteria are randomly assigned 1:1 to receive one of the following IP-BTP treatments:
  1. Fentanyl pectin nasal spray (FPNS)
  2. Physician choice-Usual Care (PC-UC)
  Interventions: Drug: Physician choice-Usual care (PC-UC)

INTERVENTIONS:
Drug: Fentanyl pectin nasal spray (FPNS) — The first dose of FPNS will be 100 mcg dose. It will be increased until 800 mcg dose.
  Arms: PecFent nasal spray
Drug: Physician choice-Usual care (PC-UC) — The PC-UC will be started at a dose according to the physician choice. If this dose of PC-UC is effective on pain control, at the following meal the patient will take the same dose of PC-UC.
  If the dose of PC-UC results non effective on pain control, at the following meal the patient will take an increased dose of the same PC-UC drug or change the PC-UC drug, according to the physician choice.
  Other Names: PC-UC is any drug used in clinical use for treating IP-BTP
  Arms: Physician choice-Usual Care (PC-UC)

SUMMARY:
The primary objective of the present phase IIIb study is to assess the efficacy of FPNS compared with Physician Choice-Usual Care (PC-UC) in the reduction of swallowing predictable BTP in head and neck cancer patients undergoing radiotherapy with or without chemotherapy.

DETAILED DESCRIPTION:
Population: In and out patients with head and neck cancer undergoing radiotherapy, regardless of the day of the radiotherapy treatment, with or without chemotherapy and taking at least 60 mg of oral morphine daily or an equianalgesic dose of another opioid to control background pain (background pain controlled is defined as NRS <4) but with uncontrolled pain at swallowing (moderate/severe intensity: ≥ 4 on a NRS 0-10).

Study design: Patients that have signed the ICF and met inclusion and exclusion criteria are randomly assigned 1:1 to receive one of the following predictable BTP at swallowing treatments:

1. Fentanyl pectin nasal spray (FPNS)
2. Physician choice-Usual Care (PC-UC) Each patient will take the drug no more than 3 episode a day (at main meals: breakfast, lunch and dinner) for 15 episodes in total in 6 (-1, +2) consecutive days. At each episode the patients will record the pain at baseline (before drug administration), and 10, 20 30 minutes after taking FPNS or PC-UC.

At each meal, if the administered dose of FPNS or PC-UC is not adequately effective on pain control, the patient is allowed to take a rescue medication of IRMS after 30 min from FPNS or PC-UC administration.

ELIGIBILITY:
Inclusion criteria:

1. Male and female aged 18 years or over
2. Diagnosis of stage III-IV cancer of oral cavity, oropharynx, hypopharynx, larynx, salivary glands
3. Receiving radiation therapy (RT) with or without concurrent platinum based chemotherapy or cetuximab as first line treatment or as postoperative adjuvant treatment
4. Background pain controlled with at least 60 mg oral morphine daily or an equianalgesic dose of another opioid. A "background pain controlled" is defined as NRS <4
5. Uncontrolled pain during swallowing (predictable BTP at swallowing) with an intensity ≥4 on an 11-point numeric scale (0=no pain; 10=worst possible pain). This pain will have to be measured with the ingestion of a solid/liquid food (depending on the ability to swallow or less solid foods of the patient at moment)
6. Patients able to receive a nasal spray therapy
7. Willing and able to sign an informed consent form
8. Females with childbearing potential must provide a negative pregnancy test and both males and females must be using adequate contraception during the study
9. Patients with PEG or jejunostomy, if are available to take by mouth meals (solid or liquid) or just liquid in order to be compliant with the protocol.

Exclusion Criteria:

1. Patients with known metastatic disease
2. Known hypersensitivity to opioids, to Fentanyl or to drugs used in the PC-UC, and/or to study medications' formulation ingredients
3. Patients with impaired chemistry laboratory exams, assessed as routine clinical practice before radiotherapy start:

   a. Hepatic function: i. Total bilirubin > 2 times the upper-normal limit (ULN) ii. Serum transaminase > 5 times ULN b. Renal function: i. Serum creatinine concentration > 2 times ULN
4. Pregnant or breastfeeding women
5. Patients unlikely to comply with the protocol or unable to understand the nature, scope and possible consequences of the study
6. Patients planned to receive other investigational treatments during study period
7. Patients with moderate to severe respiratory impairment
8. Patients with nasogastric feeding tube
9. Patients that cannot take FPNS according to investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference in the mean intensity of predictable BTP at swallowing from the baseline to 20 minutes after taking FPNS/PC-UC (PID20). | up to 6 (-1,+2) days

SECONDARY OUTCOMES:
The difference in the mean intensity of predictable BTP at swallowing from the baseline to 10 and 30 minutes after taking FPNS/PC-UC. | up to 6 (-1,+2) days
Time to reach the maximal pain reduction after administration of FPNS/PC-UC (evaluation of reduction in pain intensity score at each time point: 10,20,30 min after administration of FPNS or PC-UC) | up to 6 (-1,+2) days
Patient's swallowing pain relief will be measured at the end of the study period through the 5-points numeric scale (0=none; 4=complete). | end of study
Clinically meaningful pain reduction will be analyzed by assessing percentages of episodes with ≥ 2 point reductions after drug treatment versus baseline and after FPNS versus PC-UC | up to 6 (-1,+2) days
Administration of rescue medication (dose and frequency) | up to 6 (-1,+2) days
Patient's dysphagia assessment. An evaluation of dysphagia by MDADI questionnaire will be performed at baseline and at the end of the study period. | day 1 and end of study
Safety and tolerability | up to 6 (-1,+2) days

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Licitra, MD, Principal Investigator — Fondazione IRCCS - Istituto Nazionale Tumori - Milano (Italy)
Locations (25):
- Italy (25):
  - Ospedale Bellaria, Bologna, Bologna
  - Azienda Ospedaliera "Spedali civili" di Brescia, Brescia, Brescia
  - Ospedale Santa Croce e Carlè, Cuneo, Cuneo
  - Azienda Ospedaliera universitaria Careggi, Florence, Firenze
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.), Meldola, Forlì - Cesena
  - IRCCS AOU San Martino-IST Istituto Nazionale per la Ricerca sul Cancro, Genova, Genova
  - Ospedale Carlo Poma, Mantova, Mantova
  - Ospedale San Raffaele, Milan, Milano
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan, Milano
  - Istituto Europeo di Oncologia, Milan, Milano
  - Ospedale Niguarda Ca' Granda, Milan, Milano
  - Istituto Nazionale Tumori IRCCS - Fondazione Pascale, Napoli, Napoli
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro, Pesaro e Urbino
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - Istituto Nazionale Tumori Regina Elena, Roma, Roma
  - Policlinico Universitario Gemelli di Roma, Roma, Roma
  - Ospedale Santa Maria della Misericordia, Rovigo, Rovigo
  - Istituto per la Ricerca e la Cura del Cancro a carattere Scientifico - IRCC, Candiolo, Torino
  - Azienda Ospedaliera San luigi di Gonzaga di Orbassano, Orbassano, Torino
  - A.O. Città della Salute e della Scienza - Ospedale Dermatologico S. Lazzaro, Torino, Torino
  - Ospedale di Trento - Presidio Ospedaliero Santa Chiara, Trento, Trento
  - Azienda ULSS 9 Presidio Ospedaliero di Treviso, Treviso, Treviso
  - Azienda U.L.S.S. 12 Veneziana, Venezia Mestre, Venezia Mestre
  - Presidio Ospedaliero Mirano Azienda Ulss 13, Mirano, Venezia
  - Ospedale Sacro Cuore- dona Calabria di Negrar, Negrar, Verona